CLINICAL TRIAL: NCT00288587
Title: CP0007: Extracorporeal Ultrafiltration (UF) vs. Usual and Customary Care for Patients With Severe Heart Failure (HF)
Brief Title: Extracorporeal Ultrafiltration (UF) vs. Usual and Customary Care for Patients With Severe Heart Failure (HF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NxStage Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP0007
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-05

CONDITIONS: Heart Failure; CHF
Keywords: Heart Failure; Congestive Heart Failure; CHF
MeSH Terms: conditions — Heart Failure | interventions — Sodium Potassium Chloride Symporter Inhibitors

ARMS (2):
- Ultrafiltration (Active Comparator): Patients treated with Extracorporeal Ultrafiltration upon hospital admission for treatment of decompensated heart failure.
  Interventions: Device: NxStage System One
- Usual & Customary (Active Comparator): Patients treated with conventional diuretic therapy upon hospital admission for treatment of decompensated heart failure.
  Interventions: Drug: IV loop diuretic

INTERVENTIONS:
Drug: IV loop diuretic — Use of conventional diuretic therapy upon hospital admission for treatment of decompensated heart failure.
  Arms: Usual & Customary
Device: NxStage System One — Patients treated with Extracorporeal Ultrafiltration upon hospital admission for treatment of decompensated heart failure.
  Arms: Ultrafiltration

SUMMARY:
The purpose of this study is to assess the ability of Ultrafiltration to influence the rate of hemodynamic improvement, as measured by the decline in the pulmonary artery occlusion pressure, in patients with NYHA class III/IV Heart Failure.

DETAILED DESCRIPTION:
This study will be preformed in a specialized heart failure unit at the Cleveland Clinic Foundation (CCF) and will include both the UF-treated group and a control group receiving usual and customary care. Patients will be stratified according to renal function at the time of admission. Therapies will be guided by specific hemodynamic criteria routinely used at the study institution.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Heart Failure Unit (H-22) with NYHA class III/IV HF and pulmonary artery catheter in situ
* Left ventricular ejection fraction <40%
* Mean Pulmonary Artery Occlusion Pressure ≥20 mm Hg
* Able to give informed consent

Exclusion Criteria:

* Currently on renal replacement therapy or determined to need renal replacement therapy at the time of enrollment
* Estimated glomerular filtration rate (GFR) <15 mL/min
* Systolic blood pressure (SBP) <80 mm Hg
* Acute coronary syndrome
* Hematocrit >50%
* Malignancy other than prostrate or skin
* Chronic edematous states other than HF, including nephritic syndrome and cirrhosis
* Chronic inflammatory or infectious condition
* Pregnancy
* Previous enrollment in this study
* Expectation of need for heart transplantation or cardiac assist device within one week
* Pulmonary failure requiring intubation and mechanical ventilation
* Known or suspected hypersensitivity to dialysis membranes
* Severe aortic stenosis or regurgitation
* Severe mitral stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-10; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Hull, MD, Study Director — NxStage Medical
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Result] Hanna MA, Tang WH, Teo BW, O'Neill JO, Weinstein DM, Lau SM, Van Lente F, Starling RC, Paganini EP, Taylor DO. Extracorporeal ultrafiltration vs. conventional diuretic therapy in advanced decompensated heart failure. Congest Heart Fail. 2012 Jan-Feb;18(1):54-63. doi: 10.1111/j.1751-7133.2011.00231.x. Epub 2011 Jul 20. PMID 22277179

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual & Customary Care: Patients treated with conventional diuretic therapy upon hospital admission for the treatment of decompensated heart failure.
Period: Overall Study
Arm/Group | Ultrafiltration | Usual & Customary Care
Started | 19 | 17
Completed | 14 | 7
Not Completed | 5 | 10
Not completed — Death | 4 | 4
Not completed — Transplant | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Severe Aortic Stenosis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrafiltration | Usual & Customary Care | Total
Number analyzed (Participants) | 19 | 17 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (9.1) | 59 (15.5) | 59.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36
Glomerular Filtration Rate (GFR) [Number; unit: Participants]
  GFR >50 mL/min/1.73m2 | 9 | 10 | 19
  GFR <50 mL/min/1.73m2 | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Time Required for the Pulmonary Artery Occlusion Pressure (PAOP) to be Maintained at a Value of Less Than or Equal to 18 mmHg for at Least Four Consecutive Hours (+/- 30 Minutes) During the Intervention Period.
Time Frame: 4 consecutive hours (+/- 30 minutes)
Population: Analysis was performed on the intent-to-treat group which consisted of all patients enrolled in this study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ultrafiltration | Usual & Customary Care
Number analyzed (Participants) | 19 | 17
hours | 22.0 (4.2) | 34.8 (6.7)

2. Secondary Outcome: Time to Discharge From the Heart Failure (HF) Unit, and Time to Discharge From the Hospital.
Time Frame: Time from admission to endpoint achievement
Population: The analysis population was the intent-to-treat group, represented by all patients enrolled in this study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ultrafiltration | Usual & Customary Care
Number analyzed (Participants) | 19 | 17
Days
  Time to discharge from HF unit | 3.63 (2.11) | 3.56 (1.86)
  Time to discharge from hospital | 6.98 (4.81) | 18.93 (18.9)

3. Secondary Outcome: Total Volume Removal During the Intervention Period
Time Frame: Intervention start to end.
Population: The analysis population is the intent-to-treat group which includes all patients enrolled on the study.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Ultrafiltration | Usual & Customary Care
Number analyzed (Participants) | 19 | 17
milliliters | 5215 (3406) | 2167 (2380)

4. Secondary Outcome: Volume Removal Rate.
Description: Hours of therapy required to remove 1 liter of fluid normalized to body weight.
Time Frame: Intervention start to end.
Population: The analysis population is the intent-to-treat group which includes all patients enrolled on the study.
Measure: Mean (Standard Deviation); unit: milliliters/hour/kilogram
Arm/Group | Ultrafiltration | Usual & Customary Care
Number analyzed (Participants) | 19 | 17
milliliters/hour/kilogram | 3.4 (2.6) | 0.7 (1.1)

5. Secondary Outcome: Composite Endpoint of Hospital Readmissions, Emergency Department Visits, and Deaths
Description: Number of patients experiencing at least one of the composite endpoint measures within 90 days of hospital discharge.
Time Frame: Hospital discharge to 90 days after discharge
Population: The analysis population is the intent-to-treat group which includes all patients enrolled on the study.
Measure: Number; unit: participants
Arm/Group | Ultrafiltration | Usual & Customary Care
Number analyzed (Participants) | 19 | 17
participants | 12 | 10

ADVERSE EVENTS:
Arm/Group | Ultrafiltration | Usual & Customary Care
Serious Adverse Events (participants affected / at risk) | 4/19 | 4/17
Other Adverse Events (participants affected / at risk) | 19/19 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrafiltration (N=19) | Usual & Customary Care (N=17)
Death (Cardiac reason) (Cardiac disorders) | 3 (3) | 4 (4)
Death (Infection-related) (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrafiltration (N=19) | Usual & Customary Care (N=17)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (3)
Chest Pain (Cardiac disorders) | 2 (2) | 0 (0)
Brady Arrhythmia (Cardiac disorders) | 0 (0) | 1 (2)
Claudication (Vascular disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Cramping (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever > 37.3 C (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (2) | 1 (1)
Hypoglycemic Episode (Endocrine disorders) | 1 (1) | 0 (0)
Hypotensive Episode (Renal and urinary disorders) | 3 (3) | 4 (4)
Infection (Infections and infestations) | 3 (3) | 2 (2)
Insomnia (General disorders) | 2 (2) | 0 (0)
Nausea (General disorders) | 5 (5) | 4 (4)
Other (General disorders) | 10 (18) | 7 (11)
Painful Access (Vascular disorders) | 0 (0) | 1 (1)
Worsening Heart Failure (Cardiac disorders) | 2 (2) | 6 (7)
Worsening Renal Failure (Renal and urinary disorders) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No